CLINICAL TRIAL: NCT05027139
Title: A Phase 1b/2, 2-part Open-label Study to Assess the Safety and Antitumor Activity of Zanidatamab in Combination With ALX148 in Advanced HER2-expressing Cancer
Brief Title: A Study of Zanidatamab (ZW25) With Evorpacept (ALX148) in Patients With Advanced HER2-expressing Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: ALX Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW25-204
Expanded Access: NCT04578444 (No longer available)
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: HER2-expressing Cancers
Keywords: JZP598
MeSH Terms: interventions — zanidatamab; ALX148

STUDY DESIGN:
Intervention Model Description: single-arm, open-label, multi-cohort, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanidatamab plus evorpacept (ALX148) (Experimental)
  Interventions: Drug: Zanidatamab; Drug: Evorpacept

INTERVENTIONS:
Drug: Zanidatamab — Administered intravenously (IV)
  Other Names: ZW25; JZP598; ZIIHERA®
Drug: Evorpacept — Administered IV
  Other Names: ALX148

SUMMARY:
This study is being done to find out if zanidatamab when given with evorpacept (ALX148) is safe and can treat patients with advanced (locally advanced [inoperable] and/or metastatic) human epidermal growth factor receptor 2 (HER2)-expressing cancer.

DETAILED DESCRIPTION:
Part 1 of the study will first evaluate the safety and tolerability and establish the recommended doses (RDs) of zanidatamab in combination with evorpacept (ALX148). Part 2 of the study will evaluate the anti-tumor activity of the combination of zanidatamab plus evorpacept (ALX148) at the RD levels in indication-specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced (inoperable) and/or metastatic HER2-expressing cancer based on local or central laboratory test results as follows:

  * Parts 1 and 2: HER2-positive breast cancer as defined per American Society of Clinical Oncology (ASCO)/ College of American Pathologists (CAP) guidelines
  * Parts 1 and 2: HER2-low breast cancer (defined as immunohistochemistry [IHC] 1+ or IHC 2+; AND is currently not and has never been HER2-positive per the ASCO/CAP guidelines)
  * Part 2: HER2-positive gastroesophageal adenocarcinoma as defined per the ASCO/CAP gastric cancer-specific guidelines; or other HER2-overexpressing non-breast cancers (defined as IHC 3+; or IHC 2+ and in situ hybridization [ISH]+) per the ASCO/CAP guidelines for breast cancer
* Progression after or during the most recent systemic regimen of treatment for advanced cancer. For both Part 1 and Part 2, prior therapies must have included approved agents known to confer clinical benefit.

  * Subjects with HER2-positive breast cancer who did not receive trastuzumab or pertuzumab due to medical contraindications will not be eligible for this study
  * Subjects with HER2-low breast cancer who have received prior HER2-targeted therapy (other than trastuzumab deruxtecan, which is allowed but not required) will not be eligible for this study
* Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Willingness to undergo a new biopsy to provide a tumor tissue for central laboratory testing of HER2 protein expression and gene amplification by IHC and ISH assays, respectively
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ functions
* Adequate cardiac left ventricular function, as defined by a left ventricular ejection fraction (LVEF) ≥ 50% as determined by either echocardiogram or multiple gated acquisition scan (MUGA) obtained within 4 weeks prior to first dose of study treatment

Exclusion Criteria:

* Previous allogeneic stem cell transplant
* Prior treatment with any anti-CD47 or anti-signal regulatory protein alpha (SIRPα) agent
* Prior or concurrent invasive malignancy whose natural history or treatment has, in the opinion of the investigator or medical monitor, the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Received systemic anticancer therapy within 4 weeks of starting study treatment (6 weeks for mitomycin C or nitrosoureas). Received radiotherapy within 2 weeks of the first dose of zanidatamab/evorpacept (ALX148)
* Untreated brain metastases, symptomatic brain metastases; or radiation treatment (stereotactic radiosurgery and whole brain radiation) for brain metastases within 2 weeks of start of study treatment
* Known leptomeningeal disease
* Active hepatitis
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2. (Exception: Subjects with well controlled HIV [e.g., CD4 > 350/mm3 and undetectable viral load] are eligible.)
* QTc Fridericia (QTcF) > 470 ms
* History of myocardial infarction or unstable angina within 6 months prior to enrollment, troponin levels consistent with myocardial infarction, or clinically significant cardiac disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure
* Acute or chronic uncontrolled pancreatitis or Child-Pugh Class C liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs; Part 1) | Up to 4 weeks
  Number of patients who experienced a DLT. DLTs include specifically defined adverse events (AEs) considered to be related to zanidatamab or evorpacept (ALX148), including combination of zanidatamab with evorpacept (ALX148)
Incidence of AEs (Part 1) | Up to 7 months
  Number of patients who experienced AEs, serious adverse events (SAEs), or adverse events of special interest (AESIs)
Incidence of clinical laboratory abnormalities (Part 1) | Up to 7 months
  Number of patients who experienced a Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0
Confirmed objective response rate (ORR)(Part 2) | Up to 2 years
  Number of patients who achieved a confirmed best overall response (BOR) of either complete response (CR) or partial response (PR) during treatment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR)(Part 2) | Up to 2 years
  Number of patients who achieved a best response of CR, PR, or stable disease (SD) during treatment per RECIST 1.1
Clinical benefit rate (CBR)(Part 2) | Up to 2 years
  Number of patients who achieved a SD for ≥ 24 weeks or a confirmed BOR of CR or PR during treatment per RECIST 1.1
Duration of response (DOR)(Part 2) | Up to 2 years
  The time from the first objective response (CR or PR) to documented progressive disease per RECIST 1.1, clinical progression, or death within 30 days of last dose of study drug (zanidatamab and/or evorpacept [ALX148]) from any cause
Progression-free survival (PFS)(Part 2) | Up to 2 years
  The time from the first dose of study treatment to the date of documented disease progression (per RECIST 1.1), clinical progression, or death from any cause
Progression-free survival 6 (PFS6)(Part 2) | Up to 6 months
  Number of patients with a PFS time ≥ 24 weeks
Overall survival (OS)(Part 2) | Up to 2 years
  The time from first dose of study treatment until death from any cause
Incidence of AEs (Part 2) | Up to 7 months
  Number of patients who experienced AEs, SAEs, or AESIs
Incidence of clinical laboratory abnormalities (Part 2) | Up to 7 months
  Number of patients who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using NCI-CTCAE, version 5.0
Maximum serum concentration of zanidatamab and evorpacept (ALX148) (Part 2) | Up to 7 months
Trough concentration of zanidatamab and evorpacept (ALX148) (Part 2) | Up to 7 months
  Minimum observed serum concentration (trough)
Incidence of anti-drug antibodies (ADAs)(Part 2) | Up to 7 months
  Number of patients who develop ADAs

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - UC San Diego - Moores Cancer Center, La Jolla, California
  - UCLA Department of Medicine Hematology/Oncology, Los Angeles, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Astera Cancer Care, East Brunswick, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing